CLINICAL TRIAL: NCT05287594
Title: Feasibility of a Train-the-Trainer Delivered Exercise Intervention in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-2522
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Firefighter; High Intensity Interval Training
Keywords: Firefighter; Train-the-Trainer; High intensity interval training; Neuromuscular warm-up; Fire and Rescue Personnel
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Two group design where 40 firefighters are cluster randomized (3:2 ratio) into a TRAINER or waitlist control group. There will be 6 trainers who will lead the TRAINER condition. All participants in the TRAINER group and following the intervention in the waitlist control group will receive the same integrated exercise program, led by a peer-trainer, including a neuromuscular warm-up and high intensity interval training at their respective fire stations 2 times per week for 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAINER (Experimental): The TRAINER group will receive an integrated exercise program, led by a peer-trainer, including a neuromuscular warm-up and high intensity interval training at their respective fire stations 2 times per week for 6 weeks.
  Interventions: Behavioral: Integrated Exercise Program
- Waitlist Control (No Intervention): The waitlist control group will not receive training during the course of the study, but will be offered the opportunity to receive the integrated exercise program after the study ends.

INTERVENTIONS:
Behavioral: Integrated Exercise Program — Neuromuscular warm-up: Each participant will perform a series of dynamic stretches, core stability, balance, and medicine ball exercises. The dynamic stretches include 8 repetitions of 6 stretches targeting the hip and thigh musculature, followed by 3 core stability isometric exercises (curl-up, side bridge, and bird dog). Participants will then perform 2 sets (per leg) of hop-to-stabilization (with a reach) balance exercises, followed by 3 separate medicine ball exercises emphasizing explosive full-body movements.
  High Intensity Interval Training (HIIT): HIIT will include a series of high intensity exercise bouts on a stationary bike that includes a 1:1 work-to-rest ratio. Training intensity will be determined from the peak power output obtained during the baseline VO2 peak assessment and progressively increased by the number of bouts and intensity. The number of work bouts will increase from 5 to 8 bouts and the intensity will increase from 90 to 110% of peak power output.
  Other Names: Neuromuscular warm-up; High intensity interval training; HIIT
  Arms: TRAINER

SUMMARY:
Purpose: To collect and report feasibility data for conducting a future cluster randomized trial to evaluate the efficacy of a TRAINER delivered integrated exercise program in career firefighters, and to determine intervention fidelity and preliminary effects of a TRAINER delivered integrated exercise program in career firefighters.

Participants: 52 career firefighters 18 - 60 years old (40 trainees, 6 trainers, 6 administrators).

Procedures (methods): Enrolled fire stations will be randomly assigned (3:2 allocation ratio) to a TRAINER or wait-list control (CON) group, stratified by city, using computer-generated random numbers. All enrolled firefighters will undergo a series of assessments at baseline (week 0) and post-testing (week 7) following the TRAINER delivered 6-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent prior to any study procedures are performed
* Medically cleared for fire suppression duties
* A career firefighter from a local department (Carrboro, Chapel Hill, and Durham)

Exclusion Criteria:

* Highly active firefighters, defined as performing 4 or more days/week of vigorous exercise
* Pregnancy
* Recent injury preventing their participation in the exercise routine
* Involved in an active workers' compensation or personal injury case

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Number of Firefighters and Fire Stations Recruited to the Study (Feasibility) | Within 14 months
  To demonstrate the feasibility of an integrated exercise program. Feasibility will be defined as recruitment of 40 firefighters and the number of fire stations (out of 26 potential) to the study within 14 months.
Percentage of Firefighters Retained (Feasibility) | Week 7 (post-intervention)
  To demonstrate the feasibility of an integrated exercise program. Retention will be determined from the percentage of firefighters retained at post-testing. Retention of 80% or higher will be considered good feasibility.
Percentage of Sessions Attended (Feasibility) | Week 7 (post-intervention)
  To demonstrate the feasibility of an integrated exercise program. Adherence will be determined from the percentage of sessions attended out of total (12) sessions. Adherence of 80% or higher will be considered good feasibility.
Qualitative Summaries of Participant Experience in Semi-Structured Interviews (Acceptability) | Week 7 (post-intervention)
  Acceptability will be assessed by semi-structured interviews with the firefighters, peer-trainers, and departmental administration (e.g. fire chiefs). Qualitative summaries for intrapersonal, interpersonal, and organizational constructs will be reported.

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness as measured by VO2 peak during cycle ergometry | Baseline (i.e., pre-intervention), 7 weeks (i.e., post-intervention)
  Cardiorespiratory fitness will be measured by peak oxygen consumption (VO2 peak). All participants will perform a cycling ergometer test with respiratory gases continuously monitored with open-circuit spirometry (True One 2400®, Parvo-Medics, Inc., Provo, UT). Data will be averaged over 15-second intervals, with the highest 15-second oxygen consumption recorded as the VO2 peak.
Change in body composition as measured by % body fat from a 4-compartment model | Baseline (i.e., pre-intervention), 7 weeks (i.e., post-intervention)
  Body composition will be evaluated to determine the effects of the intervention on % body fat. Dual-energy x-ray absorptiometry (DXA;General Electric Lunar iDXA, Chicago, IL) and bioelectrical impedance spectroscopy (BIS; ImpediMed SFB7, Queensland, AU) will be used to determine a gold-standard DXA-derived four-compartment model of % body fat.
Change in explosive muscle strength as measured by dynamometry | Baseline (i.e., pre-intervention), 7 weeks (i.e., post-intervention)
  All participants will perform a rapid and maximal isometric muscle action on a calibrated isokinetic dynamometer (CSMi, Stoughton, MA) against a padded and stiff lever arm for 3-4 seconds. The peak rate of torque development will be determined from the peak of the first derivative of the torque-time curve.
Change in low-back muscular endurance as measured by a modified Biering-Sorensen test | Baseline (i.e., pre-intervention), 7 weeks (i.e., post-intervention)
  Low-back muscular endurance (time to task failure) will be examined using a modified version of the Biering-Sorensen test, using a variable angle Roman chair (Powerlift, Jefferson, IA).
Change in balance as measured by a modified star excursion balance test | Baseline (i.e., pre-intervention), 7 weeks (i.e., post-intervention)
  Balance will be determined by using a modified star excursion balance test. Following a familiarization, participants will reach with their free limb as far as possible in the anterior, posterolateral, and posteromedial direction relative to the stance leg. Scores will be normalized to leg length.
Fidelity of the neuromuscular warm-up as measured by a rubric across sessions at Week 2 | 2 weeks (i.e., beginning of intervention following train-the-trainer completion)
  The fidelity of the neuromuscular warm-up will be examined using a scoring rubric. The rubric evaluates the leadership abilities of the trainers and the execution of the exercises by the firefighters. Each item is scored 1 to 5 with 1 indicating no correctness and 5 indicating complete correctness. Items will be summed for a total score. Higher values mean higher fidelity.
Fidelity of the neuromuscular warm-up as measured by a rubric across sessions at Week 6 | 6 weeks (i.e., one of last 2 sessions)
  The fidelity of the neuromuscular warm-up will be examined using a scoring rubric. The rubric evaluates the leadership abilities of the trainers and the execution of the exercises by the firefighters. Each item is scored 1 to 5 with 1 indicating no correctness and 5 indicating complete correctness. Items will be summed for a total score. Higher values mean higher fidelity.
Fidelity of the HIIT protocol as measured by rate of peak power output across sessions at Week 2 | 2 weeks (i.e., beginning of intervention following train-the-trainer completion)
  Fidelity will be assessed to ensure participant adherence to the intervention protocol in each session. The fidelity of the HIIT protocol will be examined by recording the prescribed peak power output (90-110%) during the training session. Training intensity will be established from a percentage of the baseline peak power output (Watts) achieved during the VO2 peak test. Higher fidelity is indicated as the percent power output more closely approaches the prescribed power output percentage.
Fidelity of the HIIT protocol as measured by rate of peak power output across sessions at Week 6 | 6 weeks (i.e., one of last 2 sessions)
  Fidelity will be assessed to ensure participant adherence to the intervention protocol in each session. The fidelity of the HIIT protocol will be examined by recording the prescribed peak power output (90-110%) during the training session. Training intensity will be established from a percentage of the baseline peak power output (Watts) achieved during the VO2 peak test. Higher fidelity is indicated as the percent power output more closely approaches the prescribed power output percentage.
Change in physical activity as measured by the International Physical Activity Questionnaire-Short Form | Baseline (i.e., pre-intervention), 7 weeks (i.e., post-intervention)
  Physical activity will be examined using the validated 7-day recall International Physical Activity Questionnaire-Short Form. Higher scores represent greater total metabolic equivalent of task (MET) minutes of physical activity per week based on the following estimates: 3.3 MET units for walking, 4.4 MET units for moderate activity, 8 MET units for vigorous activity. Total MET minutes of physical activity is calculated from the questionnaire using the following calculation:
  Total MET-min/week = (Walk METs*min*days) + (Mod METs*min*days) + Vig METs*min*days)
  The study will test whether there is a BASELINE-to-POST increase in total scores on the International Physical Activity Questionnaire-Short Form (units: MET minutes/week) for the TRAINER group relative to the waitlist control group. The outcome for each group is computed as the main of the difference of the POST score minus the BASELINE score.
Change in nutrition as measured by the Rapid Eating Assessment for Participants-Short Form | Baseline (i.e., pre-intervention), 7 weeks (i.e., post-intervention)
  Nutritional habits will be examined using the validated Rapid Eating Assessment for Participants-Short Form. Responses of 'usually/often' receives 1 point, 'sometimes' receives 2 points, and 'rarely/never or does not apply to me' receives 3 points. Possible scores ranged from 13 to 39 with a higher score indicating better nutritional habits. The study will test whether there is a BASELINE-to-POST increase in total scores on the Rapid Eating Assessment for Participants-Short Form for the TRAINER group relative to the waitlist control group. The outcome for each group is computed as the main of the difference of the POST score minus the BASELINE score.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ryan, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator with IRB, IEC, or REB approval and an executed data use agreement with UNC

DOCUMENTS (1):
  • Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT05287594/ICF_000.pdf